CLINICAL TRIAL: NCT02282098
Title: Targeting Inflammation in Atrial Fibrillation to Prevent Ischemic Stroke: A Feasibility Study Evaluating the Effect of Colchicine on D-dimer and Hs-CRP in Anticoagulated Patients With Atrial Fibrillation
Brief Title: Colchicine in Atrial Fibrillation to Prevent Stroke
Acronym: CIAFS-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Responsible Party: Principal Investigator, Noel Chan, PI, Population Health Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NIF-14350; NIF-14350 (Other Grant/Funding Number: Hamilton Health Science New Investigator Fund)
Record Dates: First submitted 2014-10-29; First posted 2014-11-04 (Estimated); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Atrial Fibrillation; Stroke
Keywords: Atrial fibrillation; Arrhythmias, Cardiac; Stroke; agents, anti inflammatory; D-dimer; C-reactive protein
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Arrhythmias, Cardiac | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Colchicine (Experimental): The intervention group will receive colchicine 0.6 mg twice daily orally for 3 months
  Interventions: Drug: Colchicine
- Placebo Colchicine (Placebo Comparator): The control group will receive colchicine placebo 0.6mg twice daily orally for 3 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colchicine — Colchicine 0.6mg twice daily
  Other Names: pms-Colchicine
  Arms: Active Colchicine
Drug: Placebo — Placebo Colchicine
  Other Names: Placebo Capsule
  Arms: Placebo Colchicine

SUMMARY:
The purpose of this study is to determine the feasibility of performing a randomized controlled trial to investigate the efficacy of an anti-inflammatory drug, colchicine, at reducing well validated markers of thrombosis (D-dimer) and inflammation (hs-CRP).

DETAILED DESCRIPTION:
Atrial fibrillation (AF), the most common cardiac arrhythmia (with a global burden of 33.5 million affected patients in 2010), is responsible for about 20% of ischemic stroke, a major cause of morbidity and mortality. Anticoagulants are very effective in reducing the risk of stroke in AF but on average 10-15% of treated patients still experience a stroke over a 10-year period and in selected elderly populations the risk is even higher. We hypothesize that thrombosis mediated by inflammation might be responsible for the residual risk of stroke, despite anticoagulant therapy and that targeting inflammation has the potential to reduce thrombosis and the risk of stroke in anticoagulated patients with AF.

ELIGIBILITY:
Inclusion Criteria:

* Patients with atrial fibrillation who has been receiving chronic anticoagulation for at least 3 months.

Exclusion Criteria:

* Contraindications to colchicine such as allergy/hypersensitivity,
* Receiving colchicine or other anti-inflammatory drugs (such as corticosteroids, methotrexate, anti-neoplastic, Interleukin 1-1b antagonist, Tumor necrosis factor-alpha inhibitor),
* Receiving food or co-medications such as strong-moderate cytochrome P450 3A4 inhibitors that will result in elevated plasma level of colchicine,
* Inflammatory disorders (SLE, Rheumatoid arthritis, connective tissue disorder) or chronic infection,
* Severe renal (eGFR< 30ml/min/1.73m2), or liver failure or liver aminotransferase (ALT/AST > 2x Upper limit of normal),
* Moderate or severe cytopenias (platelet < 100, neutrophil count < 1.5) or existing blood dyscrasia (e.g., myelodysplasia)
* Pregnant or lactating woman or woman of child bearing age no protected by reliable contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-11; Primary Completion 2020-11-17 (Actual); Study Completion 2020-11-17 (Actual)

PRIMARY OUTCOMES:
Recruitment rates | Randomization to Month 3
  Number of eligible patients successfully randomized into study per year of study.
Drop-out rates | Randomization to Month 3
  Proportion of participants withdrawing from study for any reason

SECONDARY OUTCOMES:
D-dimer | Randomization to Month 3
  Mean D-dimer level at baseline and Month 3 for each arm
hs-CRP | Randomization to Month 3
  Mean level of hs-CRP at baseline and month 3 for each arm
Proportion of patients with a clinically significant adverse event | Randomization to Month 3
  Proportion of patients with side effects such as diarrhoea, myopathy requiring drug cessation
Drug adherence | Randomization to Month 3
  Proportion of missing pill to dispensed pill at 6 weeks and month 3

CONTACTS AND LOCATIONS:
Overall Officials: Noel Chan, MD, Principal Investigator — Population Health Research Institute; John Eikelboom, MD, Principal Investigator — Population Health Research Institute
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada